CLINICAL TRIAL: NCT00994357
Title: The Effect of Real-time Continuous Glucose Monitoring on Severe Complications to Pregnancy in Women With Diabetes: a Randomised Controlled Study
Brief Title: The Effect of Real-time Continuous Glucose Monitoring on Severe Complications to Pregnancy in Women With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Anna Lilja Secher, MD, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SENSOR-01
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes; Pregnancy
Keywords: Real-time Continuous Glucose Monitoring; Macrosomia
MeSH Terms: conditions — Diabetes Mellitus | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real-time Continuous Glucose Monitoring (Experimental): Real-time Continuous Glucose Monitoring at five times for up to 6 days during pregnancy, and during delivery, in addition to standard monitoring and treatment.
  Interventions: Device: Real-time CGM
- Control group (Active Comparator): Standard monitoring and treatment of diabetic patients during pregnancy.
  Interventions: Other: Standard care

INTERVENTIONS:
Device: Real-time CGM — See previous description.
  Arms: Real-time Continuous Glucose Monitoring
Other: Standard care — See text.
  Arms: Control group

SUMMARY:
The purpose of the study is to investigate the effects of Real-time Continuous Glucose Monitoring on severe complications to pregnancy in women with diabetes.

DETAILED DESCRIPTION:
Pregnancy outcome in women with type 1 or type 2 diabetes is still significantly poorer than in the background population. The prevalence of large fat babies (LGA) is 50% in both types of diabetes, and perinatal death and preterm delivery is 4-7 times higher than in non-diabetic women. These complications are all closely related to non-optimal glycemic control in pregnancy, and improved metabolic control is crucial in our strive for improved pregnancy outcome in these patients.

In 2007, a new generation of "real-time" Continuous Glucose Monitoring (CGM) became available in Denmark. These sensors estimate tissue glucose values automatically and frequently with immediate display of the glucose level. In addition it is possible to set alarms for high and low glucose levels, and the patient can react immediately with changes in diet or insulin dose.

In this trial, 154 patients were randomized to either continuous glucose monitoring at five times in pregnancy in addition to standard care ot to unchanged standard care. The main aim is to evaluate if the use of CGM in pregnancy can reduce the prevalence of LGA from 50 to 30%, but other outcome measurements such as preterm delivery, neonatal disease, hypoglycemia, low grade inflammation and vascular dysfunction, quality of life and self- care are also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Pregestational diabetes, type 1 or type 2
* Single intrauterine pregnancy
* At least 18 years old
* Informed consent

Exclusion Criteria:

* Past gestational week 14 at inclusion
* Mental disorders
* Language barriere
* Gemelli
* Diabetic nephropathy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2009-02; Primary Completion 2011-10 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of LGA in children of diabetic women. | Obtained shortly after birth

SECONDARY OUTCOMES:
Metabolic control in terms of HbA1c, blood sugar measurements and the occurence of severe hypoglycemia in pregnant diabetic patients. | During pregnancy
Quality of life, locus of control and anxiety and depression scores in pregnant diabetic patients. | During pregnancy
Neonatal disease such as neonatal hypoglycemia, respiratory distress and the occurrence of malformations in children of diabetic mothers. | Shortly after birth
The occurrence of low grade inflammation and endothelial dysfunction in pregnant women with diabetes. | During pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth R Mathiesen, M.D., Study Chair — Center for Pregnant Women with Diabetes, Copenhagen University Hospital

REFERENCES:
- [Derived] Cordua S, Secher AL, Ringholm L, Damm P, Mathiesen ER. Real-time continuous glucose monitoring during labour and delivery in women with Type 1 diabetes - observations from a randomized controlled trial. Diabet Med. 2013 Nov;30(11):1374-81. doi: 10.1111/dme.12246. Epub 2013 Jul 26. PMID 23758126
- [Derived] Secher AL, Ringholm L, Andersen HU, Damm P, Mathiesen ER. The effect of real-time continuous glucose monitoring in pregnant women with diabetes: a randomized controlled trial. Diabetes Care. 2013 Jul;36(7):1877-83. doi: 10.2337/dc12-2360. Epub 2013 Jan 24. PMID 23349548